CLINICAL TRIAL: NCT03151954
Title: Yap, the Nuclear Target of Hippo Signaling, Regulates Nasal Epithelium Stem Cells Aberrant Proliferation and Differentiation in Nasal Polyps
Brief Title: The Activation of Hippo Pathway in Nasal Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Deng Huiyi, Postgraduate, Head of Otolaryngology, Principal Investigator, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSFC-H1301
Record Dates: First submitted 2017-04-21; First posted 2017-05-12 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Nasal Polyps
Keywords: nasal epithelium stem cells; Hippo-YAP pathway; proliferation; differentiation
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nasal polyps (Experimental): 1. Explore the degree of abnormal proliferation in NESCs,and analyze the relationship between the proliferation and the activation of hippo-YAP pathway,then explore the levels of LPS and Th2/17 cytokines in nasal polyps,and the relation between cytokines and the activation of hippo-YAP pathway through Immunohistochemistry and Immunofluorescence （P63、Ki67、YAP、LATS1/2 and MST1/2），as well as Western Blot and the Flow cytometry.
  2. Explore if the LPS and LPS and Th2/17 cytokines, as well as the epidermal growth factors can effect the hippo-YAP pathway of NESCs through cell culture, Western Blot and Real time PCR,and test the YAP expression and location through Immunohistochemistry.
  3. Explore that how the hippo-YAP effect the proliferation and differentiation of NESCs through cell transfection;
  4. Explore the regulation of hippo-YAP pathway in NESCs.
  Interventions: Procedure: functional endonasal sinus surgery
- inferior turbinate (Placebo Comparator): Compared with nasal polyps,explore the levels of LPS and Th2/17 cytokines in nasal polyps,and the relation between cytokines and the activation of hippo-YAP pathway through Immunohistochemistry and Immunofluorescence（P63、Ki67、YAP、LATS1/2 and MST1/2），as well as Western Blot and the Flow cytometry.
  Interventions: Procedure: nasal septal construction

INTERVENTIONS:
Procedure: functional endonasal sinus surgery — collect nasal polyps from patients
  Other Names: FESS
  Arms: nasal polyps
Procedure: nasal septal construction — collect inferior turbinates from patients as control arm
  Arms: inferior turbinate

SUMMARY:
Hippo-YAP pathway is a newly discovered pathway controlling the growth, and plays important roles in the regulation of stem cell function and tissue regeneration. Previously we found that a higher expression of YAP in NP, and LPS was able to activate the hippo-YAP pathway in NESCs. Thus, we hypothesize that the aberrant proliferation and differentiation of NESCs could be regulated via the hippo-YAP pathway.

DETAILED DESCRIPTION:
Studies have shown that the development of nasal polyps (NP) are closely related to the epithelial remodeling.The investigators have shown that nasal epithelial stem cells(NESCs) derived from NP had reduced growth and proliferation dynamics in vitro culture,and differentiated into ciliated cells with impaired cilia architecture and ciliogenesis.Further studies demonstrated that NESCs were involved in the aberrant damage repair process of the epithelial remodeling in NP.Hippo-YAP pathway is a newly discovered pathway controlling the growth,and plays important roles in the regulation of stem cell function and tissue regeneration.Previously the investigators found that a higher expression of YAP in NP,and LPS was able to activate the hippo-YAP pathway in NESCs.Thus,the investigators hypothesize that the aberrant proliferation and differentiation of NESCs could be regulated via the hippo-YAP pathway,which may result in the epithelial remodeling.In this study,the investigators intend to investigate the mechanism of the hippo-YAP pathway in regulating aberrant proliferation and differentiation of NESCs and explore its upstream signaling and downstream target genes,using the NESCs gas-liquid interface culture system,and a silencing and overexpression of the hippo-YAP pathway component strategy.The investigators aim to unravel the effect and mechanism of the hippo-YAP pathway in the epithelial remodeling of NP,providing new targets and strategy for the improvement or reversal of NP epithelial remodeling.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of nasal polyps or deviation of nasal septum based on CT
* Must be able to withstand surgery
* At least 18 years old
* A sufficient level of education to understand study procedures and be able to communicate with site personnel and adhere to the follow-up;
* Accepted informed consent verbally and in writing

Exclusion Criteria:

* The Poor Health
* Be allergic to anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
location of YAP in tissues | through study completion, an average of 2 years
  through Immunohistochemistry
protein expression level of YAP in tissues | through study completion, an average of 2 years
  through western blot

SECONDARY OUTCOMES:
expression level of Th1 cytokines in the tissues | through study completion, an average of 2 years
  through Flow cytometry
expression level of Th17 cytokines in the tissues | through study completion, an average of 2 years
  through Flow cytometry
activation of hippo-YAP in NSECs on protein aspect | through study completion, an average of 2 years
  Western Blot
activation of hippo-YAP in NSECs | through study completion, an average of 2 years
  Flow cytometry
activation of hippo-YAP in NSECs on gene aspect | through study completion, an average of 2 years
  quantitive real time PCR

CONTACTS AND LOCATIONS:
Locations (1):
- ThirdSunYatSen, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided